CLINICAL TRIAL: NCT05350072
Title: A Randomized, Double-blind, Placebo Controlled, 2-arm Multicenter Phase 3 Study to Assess the Efficacy and Safety of Ianalumab in Patients With Active Sjogren's Syndrome (NEPTUNUS-1)
Brief Title: Two-arm Study to Assess Efficacy and Safety of Ianalumab (VAY736) in Patients With Active Sjogren's Syndrome
Acronym: NEPTUNUS-1
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CVAY736A2301; 2024-511069-12-00 (Registry Identifier: EU CT NUMBER)
Record Dates: First submitted 2022-04-07; First posted 2022-04-27 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Sjogren Syndrome
Keywords: Sjogren's syndrome; B-cell depleting; BAFF-R; VAY736; ianalumab; NEPTUNUS
MeSH Terms: conditions — Sjogren's Syndrome | interventions — ianalumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, investigators, investigator staff, persons performing the assessments and Novartis Clinical Trial Team will remain blinded to the identity of the treatment from the time of randomization until the final database lock.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): ianalumab
  Interventions: Biological: VAY736
- Arm B (Placebo Comparator): placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: VAY736 — ianalumab s.c.
  Arms: Arm A
Other: Placebo — placebo s.c.
  Arms: Arm B

SUMMARY:
A randomized, double-blind, placebo controlled, 2-arm multicenter phase 3 study to assess the efficacy and safety of ianalumab in patients with active Sjogren's syndrome (NEPTUNUS-1)

DETAILED DESCRIPTION:
Two-arm study of the clinical efficacy, safety and tolerability of ianalumab (VAY736) in patients with active Sjogren's syndrome. The purpose of the study is to demonstrate the clinical efficacy, safety and tolerability of ianalumab (VAY736) administered subcutaneously (s.c.) monthly compared to placebo in patients with active Sjogren's syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent must be obtained prior to participation in the study
* Women and men ≥ 18 years of age
* Classification of Sjögren's syndrome according to the ACR/EULAR 2016 criteria
* Time since diagnosis of Sjögren's of ≤ 7.5 years at screening
* Positive anti-Ro/SSA antibody at screening

  * Patients negative for anti-Ro/SSA antibody are eligible, if they have a positive salivary gland biopsy confirmed by central expert review
  * Enrollment of anti-Ro/SSA-negative patients will be limited up to ≤10% of the study population
* Screening ESSDAI score of ≥ 5 within the following 8 domains: constitutional, lymphadenopathy, glandular, articular, cutaneous, renal, hematological and biologic.
* Stimulated whole salivary flow (sSF) rate of ≥ 0.05 mL/min at screening
* Ability to communicate well with the Investigator, understand and agree to comply with the requirements of the study
* Patients taking hydroxychloroquine (≤ 400 mg/day), methotrexate (≤ 25 mg/week) or azathioprine (≤ 150 mg/day) alone or in combination, are allowed to continue their medication, and must have been on a stable dose for at least 30 days prior to randomization.
* Patients taking systemic corticosteroids have to be on a stable dose of ≤ 10 mg/day predniso(lo)ne or equivalent for at least 30 days before randomization.
* Patients taking

  * disease-modifying antirheumatic drugs (DMARDs) other than specifically allowed by protocol
  * the following Traditional Chinese Medicines: Total glucoside of peony (TGP) or Tripterium glycosides (TG) must discontinue these medications at least 30 days prior to randomization, except for leflunomide, which has to be discontinued for 8 weeks prior to randomization unless a cholestyramine wash-out has been performed.

Exclusion Criteria:

* Presence of another autoimmune rheumatic disease that is active and constitutes the principal illness
* Use of other investigational drugs within 5 half-lives of enrollment, or within 30 days or until the expected pharmacodynamic effect has returned to baseline, whichever is longer3. Prior treatment with ianalumab
* Prior use of a B-cell depleting therapy other than ianalumab within 36 weeks prior to randomization or as long as B-cell count is less than the lower limit of normal or baseline value prior to receipt of previous B cell-depleting therapy (whichever is lower)
* Prior treatment with any of the following:

  1. Within 24 weeks prior to randomization: iscalimab (anti CD-40 mAb), belimumab , abatacept, anti-tumor necrosis factor alpha biologic agents, immunoglobulins plasmapheresis;
  2. Within 12 weeks prior to randomization: i.v. or oral cyclophosphamide and mycophenolate mofetil, i.v. or oral cyclosporine A or any other immunosuppressants (e.g., JAK inhibitors or other kinase inhibitors) unless explicitly allowed by protocol
* Use of corticosteroids (predniso(lo)ne or equivalent corticosteroid) at dose >10 mg/day
* Any one of the following laboratory values at screening:

  * Hemoglobin levels < 8.0 g/dL
  * White blood cells (WBC) count < 2.0 x 10E3/µL
  * Platelet count < 80 x 10E3/µL
  * Absolute neutrophil count (ANC) < 0.8 x 10E3/µL
* Active viral, bacterial or other infections requiring systemic treatment at the time of screening or randomization, or history of recurrent clinically significant infection or of recurrent bacterial infections with encapsulated organisms
* History of hypersensitivity to any of the study drugs or its excipients or to drugs of similar chemical classes (e.g., mAb of IgG1 class) or to any of the constituents of the study drug formulation (sucrose, L-histidine hydrochloride/ L-histidine, polysorbate 20)
* History of major organ, hematopoietic stem cell or bone marrow transplant
* Required regular use of medications known to cause dry mouth/eyes as a regular and major side effect, and which have not been on a stable dose for at least 30 days prior to Screening, or any anticipated change in the treatment regimen during the course of the study
* Use of topical ocular prescription medications (excluding artificial tears, gels, lubricants) that have not been on a stable dose for at least 90 days prior to randomization, or any anticipated change in the treatment regimen during the course of the study
* Receipt of live/attenuated vaccine within a 4-week period prior to randomization
* History of primary or secondary immunodeficiency, including a positive human immunodeficiency virus (HIV) test result
* History of malignancy of any organ system (other than localized basal cell carcinoma of the skin or in situ cervical cancer or Sjögren's related lymphoma), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
* History of sarcoidosis
* Any surgical, medical (e.g., uncontrolled hypertension, heart failure or diabetes mellitus), psychiatric or additional physical condition that the Investigator feels may jeopardize the patient in case of participation in this study
* Chronic infection with hepatitis B (HBV) or hepatitis C (HCV) virus. Positive serology for hepatitis B surface antigen (HBsAg) excludes the subject.

  * HBsAg negative subjects who are hepatitis B core antibody (HBcAb) positive are also excluded unless all of the following criteria are met:

    1. HBV DNA is negative
    2. hepatitis B monitoring is implemented - in these subjects, monthly testing of HBsAg and HBV DNA must be performed while on study treatment and at least every 12 weeks after end of treatment for the entire duration of safety follow-up.
    3. Antiviral prophylaxis must be implemented before the first administration of the study treatment, and continued up to 12 months after the end of study treatment. If antiviral therapy cannot be given or if the patient is not willing to comply with the antiviral treatment requirement, the patient is not eligible for the study.
  * Hepatitis C: patients with positive hepatitis C antibody and HCV-RNA at screening are excluded. Chronic hepatitis C patients who have completed HCV anti-viral treatment must be HCV-RNA negative at least 12 weeks after treatment before randomization to be eligible. Cases of spontaneous HCV clearance should be discussed with sponsor before enrollment.
* Evidence of active tuberculosis (TB) infection is exclusionary. Patients with previously treated TB and previously treated or newly diagnosed latent TB may be eligible.
* Pregnant or nursing (lactating) women.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception while on study treatment and for 6 months after stopping of investigational medication.
* Patients with a known history of non-compliance to medication, or who were unable or unwilling to complete PRO questionnaires, or who are unable or unwilling to use the device for collection of PROs.
* United States (and other countries, if locally required): Sexually active males, unless they agree to use barrier protection during intercourse with a woman of childbearing potential, while taking study treatment. As condom use alone has a reported failure rate exceeding 1% per year, it is recommended that female partners of male study participants use a second method of birth control. Although ianalumab is not teratogenic and/or genotoxic, and not transferred to semen, male contraception is required, as requested by FDA.

Globally, for all sexually active males, contraception should be used in accordance with locally approved prescribing information of concomitant medications administered.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2022-07-28 (Actual); Primary Completion 2025-05-07 (Actual); Study Completion 2027-05-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in EULAR Sjogren Syndrome Disease Activity Index (ESSDAI) score at Week 48 as compared to placebo | 48 weeks
  Efficacy (Plan A: US and US reference countries and Plan B: EU, China, other non-US Regions and EU reference countries)
  Dose response measured by change multi-dimensional disease activity as assessed by the physician. Score range is 0-123. Higher scores on the EULAR Sjogren's Syndrome Disease Activity Index (ESSDAI) scale are associated with poorer health states A negative change from baseline indicates improvement in disease status.

SECONDARY OUTCOMES:
Achieving ESSDAI response at Week 48 | 48 weeks
  Efficacy (Plan A and B)
  Dose response measured by change multi-dimensional disease activity as assessed by the physician. Score range is 0-123. Higher scores on the EULAR Sjogren's Syndrome Disease Activity Index (ESSDAI) scale are associated with poorer health states A negative change from baseline indicates improvement in disease status.
Achieving ESSDAI score <5 at Week 48 | 48 weeks
  Efficacy (Plan A and B)
  Dose response measured by change multi-dimensional disease activity as assessed by the physician. Score range is 0-123. Higher scores on the EULAR Sjogren's Syndrome Disease Activity Index (ESSDAI) scale are associated with poorer health states A negative change from baseline indicates improvement in disease status.
Achieving ESSDAI response at Week 24 | 24 weeks
  Efficacy (Plan A and B)
  Dose response measured by change multi-dimensional disease activity as assessed by the physician. Score range is 0-123. Higher scores on the EULAR Sjogren's Syndrome Disease Activity Index (ESSDAI) scale are associated with poorer health states A negative change from baseline indicates improvement in disease status.
Achieving SSSD response at Week 48 | 48 weeks
  Efficacy (Plan B)
  The Sjogrens Syndrome Symptom Diary (SSSD) is questionnaire consists of five (six for females) questions about symptoms of Sjögren's syndrome, each question given a score of 0-10 (0=no symptoms, 10=worst possible symptoms) where patient choose the one response that best describes how severe the symptom was at its worst in the PAST 24 HOURS. It includes six symptom items (eye dryness, mouth dryness, skin dryness, physical fatigue, muscle and/or joint pain, genital dryness), and applies a recall period of 24 hrs. The aim of the SSSD is to establish patient reported endpoints for the treatment of Sjogrens syndrome. Participants will complete the diary daily for 7 days prior to the scheduled dosing.
Change from baseline in stimulated whole salivary flow rate at Week 48 | 48 weeks
  Efficacy (Plan A and B)
Change from baseline in Physician's Global Assessment (PhGA) of disease activity at Week 48 | 48 weeks
  Efficacy (Plan A and B)
Change from baseline in Patient's Global Assessment (PaGA) of disease activity at Week 48 | 48 weeks
  Efficacy (Plan A and B)
Change from baseline in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) score at Week 48 | 48 weeks
  Efficacy (Plan A and B)
Achieving EULAR Sjögren Syndrome Patient Reported Index (ESSPRI) response at Week 48 | 48 weeks
  Efficacy (Plan B)

OTHER OUTCOMES:
Incidence of Treatment Emergent Adverse Event (TEAEs)/Serious Adverse Events (SAEs) upto the end of the study | through study completion upto 2 years
  Safety (Plan A and B)
Incidence of anti-ianalumab antibodies in serum Anti Drug Antibody (ADA) assay) up to end of study | through study completion up to 2 years
  Immunogenicity (Plan A and B)
Ianalumab concentration in serum during the treatment (example Ctrough) and follow-up (up to end of study) | through study completion up to 2 years
  Pharmacokinetics (Plan A and B)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (72):
- United States (14):
  - Medvin Clinical Research, Van Nuys, California
  - West Broward Rheumatology Associates Inc, Tamarac, Florida
  - Indiana Univ School of Dentistry, Indianapolis, Indiana
  - Ochsner Health System, Baton Rouge, Louisiana
  - The John Hopkins Jerome L Greene Sjogren, Baltimore, Maryland
  - Winthrop University Hospital, Mineola, New York
  - Carolina Arthritis Associates, Wilmington, North Carolina
  - STAT Research Inc, Dayton, Ohio
  - Altoona Center for Clin Res, Duncansville, Pennsylvania
  - Prisma Health, Columbia, South Carolina
  - Precision Comprehensive Research, Colleyville, Texas
  - Metroplex Clinical Research, Dallas, Texas
  - Baylor College Of Medicine, Houston, Texas
  - Houston Rheumatology & Arthrit, Katy, Texas
- Austria (2):
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Stockerau
- Novartis Investigative Site, Leuven, Belgium
- Brazil (4):
  - Novartis Investigative Site, Vitória, Espírito Santo
  - Novartis Investigative Site, Juiz de Fora, Minas Gerais
  - Novartis Investigative Site, Ribeirão Preto, São Paulo
  - Novartis Investigative Site, São Paulo
- Novartis Investigative Site, Santiago, Santiago Metropolitan, Chile
- China (11):
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Shenzhen, Guangdong
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Baotou, Inner Mongolia
  - Novartis Investigative Site, Hohhot, Inner Mongolia
  - Novartis Investigative Site, Nanchang, Jiangxi
  - Novartis Investigative Site, Shenyang, Liaoning
  - Novartis Investigative Site, Linyi, Shandong
  - Novartis Investigative Site, Taiyuan, Shanxi
  - Novartis Investigative Site, Xian, Shanxi
  - Novartis Investigative Site, Beijing
- Czechia (3):
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Prague
  - Novartis Investigative Site, Uherské Hradiště
- France (6):
  - Novartis Investigative Site, Caen
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Saint-Priest-en-Jarez
- Germany (6):
  - Novartis Investigative Site, Freiburg im Breisgau, Baden-Wurttemberg
  - Novartis Investigative Site, Würzburg, Bavaria
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Gommern
  - Novartis Investigative Site, Ludwigshafen
- Guatemala (2):
  - Novartis Investigative Site, Guatemala City
  - Novartis Investigative Site, Quetzaltenango
- Novartis Investigative Site, Vilnius, Lithuania
- Mexico (2):
  - Novartis Investigative Site, Guadalajara, Jalisco
  - Novartis Investigative Site, Mexico City, Mexico City
- Poland (4):
  - Novartis Investigative Site, Wroclaw, Lower Silesian Voivodeship
  - Novartis Investigative Site, Bydgoszcz
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Lublin
- Portugal (3):
  - Novartis Investigative Site, Braga
  - Novartis Investigative Site, Guarda
  - Novartis Investigative Site, Lisbon
- Novartis Investigative Site, Singapore, Singapore
- South Korea (2):
  - Novartis Investigative Site, Gwangju
  - Novartis Investigative Site, Seoul
- Spain (5):
  - Novartis Investigative Site, Badalona, Barcelona
  - Novartis Investigative Site, Sabadell, Barcelona
  - Novartis Investigative Site, Bilbao, Bizkaia
  - Novartis Investigative Site, A Coruña
  - Novartis Investigative Site, Madrid
- Turkey (Türkiye) (4):
  - Novartis Investigative Site, Ankara, Bilkent Cankaya
  - Novartis Investigative Site, Ankara, Sihhiye-Altindag
  - Novartis Investigative Site, Ankara, Yenimahalle
  - Novartis Investigative Site, Kocaeli

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com